CLINICAL TRIAL: NCT05374824
Title: Comparative Effectiveness of Palliative Surgery Versus Additional Anti-Seizure Medications for Lennox-Gastaut Syndrome - PCORI
Brief Title: Comparative Effectiveness of Palliative Surgery Versus Additional Anti-Seizure Medications for Lennox-Gastaut Syndrome
Acronym: SOM-L
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Nationwide Children's Hospital (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Pittsburgh (Other); Seattle Children's Hospital (Other); St. Louis Children's Hospital (Other); University of Cincinnati (Other); Nemours Children's Health System (Other); Stanford University (Other); Monroe Carell Jr. Children's Hospital at Vanderbilt (Other); University of North Carolina (Other); Duke University (Other); Indiana University (Other); Johns Hopkins University (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Principal Investigator, Sandi Lam, Chief, Division of Pediatric Neurosurgery, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2021-4532; RD-2020C2-20356 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2022-05-06; First posted 2022-05-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lennox Gastaut Syndrome
Keywords: epilepsy; seizure
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lennox-Gastaut syndrome is a serious and rare form of epilepsy that begins in infancy and early childhood. Seizures and their consequences need medical attention, emergency encounters, and hospitalizations. Seizures disrupt home life for the patient and for family. Lennox-Gastaut syndrome is typically accompanied by disabilities in motor, communication, eating, and other skills needed for daily function.

Lennox-Gastaut syndrome (LGS) has no cure. Although current treatments may help reduce the number of seizures, none are expected to eliminate them entirely; these treatments are palliative. The main treatments include anti-seizure medications and some surgical approaches, including the implantation of a vagus nerve stimulator (a pacemaker-like generator implanted in the chest wall and programmed by a physician to stimulate the vagus nerve in the neck) and corpus callosotomy (cutting through the band of fibers that connect the two sides of the brain). While both types of treatment (medications and surgeries) produce some benefit by reducing how often the seizures occur, both also have some risks. All medications can, in some patients, produce moderate to severe side effects. This is true of anti-seizure medications. Most patients with LGS take several anti-seizure medications at a time. Surgeries can also have associated risks and is additionally stressful for parents and family members. Currently, there is no strong evidence to support parents and physicians in deciding which type of treatment (more medicines or surgery) will be most successful for a child with LGS, and whether one or the other approach may lessen the toll that seizures take on a child's development and ability to function.

This study has two components. It will engage a network of seven pediatric hospitals in the United States where children with Lennox-Gastaut syndrome are cared for and determine whether seizure-related emergency department visits and hospitalizations are more likely to be reduced following the use of additional medications or adding palliative surgery to existing medications. The investigators will determine whether medical versus surgical treatment is more likely to lessen some of the developmental and functional difficulties that affect patients with LGS. The study will also determine whether starting therapies at a younger versus older age makes a difference.

The second component of the study will provide a description of the use of surgical versus medical treatment approaches across 18 pediatric hospitals in the United States (seven plus 11 centers). The investigators will describe how treatments differ across hospitals and over time.

The results from this study will help parents and providers make more informed choices about treatment for children with Lennox-Gastaut syndrome and will highlight areas for improvement in providing the best possible health care for this severe, lifelong disorder.

DETAILED DESCRIPTION:
Background and Significance: Lennox-Gastaut Syndrome (LGS) is a rare developmental-epileptic encephalopathy characterized by life-long refractory seizures which result in frequent utilization of emergency healthcare resources and also contribute to the severe developmental and functional impairment ubiquitously seen in affected patients. Current treatment pathways are the addition of anti-seizure medication treatment or palliative surgical procedures (including neurostimulation), both of which have strong evidence supporting their effectiveness in reducing seizure frequency, but without cures. No evidence exists about the comparative effectiveness of these two pathways. Until such evidence is developed, parents and physicians will continue to struggle with difficult and daunting decisions about whether to add anti-seizure medications or to pursue palliative surgery, and when to do so.

Study Aims: Determine the comparative effectiveness of adding palliative surgery versus adding an LGS-approved medication (Aim 1a) for decreasing utilization of seizure-related emergency health care and (Aim 1b) for limiting the impairment of functional abilities. (Aim 2) Describe the frequency and patterns of utilization of the two therapy pathways at 18 PCORnet sites for variation over time and across sites as well as by patient features - age, medical fragility, race, ethnicity, and insurance type. In addressing these aims, the study will assess and improve PCORnet infrastructure and will enhance methods for future studies of LGS and other rare epilepsies.

Study Description: (Aim 1a) Observational retrospective cohort study of emergency health-care utilization and (Aim 1b) cross sectional study of the impact of treatment pathways on functional outcomes. (Aim 2) Retrospective open cohort study of frequency and patterns (by race, ethnicity, insurance, age) of utilization of the two treatment pathways.

ELIGIBILITY:
Inclusion Criteria:

Patients with the diagnosis of Lennox Gastaut syndrome with medical records at the seven plus eleven pediatric centers

Exclusion Criteria:

Patients without Lennox Gastaut Syndrome

Max Age: 26 Years | Sex: All
Age Groups: Child, Adult
Study Population: For Aim 1a, 928 patients up to age 30 years with a chart-review validated diagnosis of Lennox-Gastaut Syndrome between 1/1/2016 and 12/31/2021 will be identified from 7 principal pediatric hospitals. For Aim 1b, a subset of half of those 928 patients (N=464) will be recruited. Analyses for Aim 2 will be based on ≥4000 patients with LGS ICD-10 codes from 18 pediatric hospitals (representing 5 PCORnet CRNs).
Sampling Method: Probability Sample
Enrollment: 4680 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Seizure-related emergency health care utilization | 2 years
  Emergency health-care utilization for Aim 1a will be defined as the frequency per year of seizure-related emergency department visits and separately seizure-related inpatient admissions in the two years postintervention (surgery or medical), with adjustment for the rate during the year prior to intervention.

SECONDARY OUTCOMES:
Parent-reported Clinical Outcome Assessments | 2 years
  Parent-reported qualitative input through descriptive assessment. The measures will be assessed once.

CONTACTS AND LOCATIONS:
Overall Officials: Sandi Lam, MD MBA, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (4):
- United States (4):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam S, Rosenman M, Dixon-Salazar T, Knupp KG, Thio LL, Abel TJ, Welch WP, Reed L, Randle SC, Garcia-Sosa R, Hauptman JS, Foster CC, Alpern ER, Zhang L, Villalba N, Carroll M, Patel AD. Comparative effectiveness of epilepsy surgery versus additional anti-seizure medications for Lennox-Gastaut syndrome: study protocol for a multicenter, mixed-methods study. Front Neurol. 2025 Jun 18;16:1569551. doi: 10.3389/fneur.2025.1569551. eCollection 2025. PMID 40606139
- See also: PCORI website — https://www.pcori.org/research-results/2021/comparing-two-treatments-children-lennox-gastaut-syndrome
- See also: Project Page — https://lgsresearch.org/